CLINICAL TRIAL: NCT02882464
Title: Evaluation of Dose-dependent Platelet-rich Fibrin Membrane Effect on Treatment of Gingival Recessions: A Randomized, Controlled, Parallel-designed Clinical Trial
Brief Title: Effect of Dose-dependent Platelet Rich Fibrin(PRF)
Acronym: PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rana Culhaoglu, Dr Dt, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/3
Record Dates: First submitted 2016-06-05; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Gingival Recession
Keywords: gingival recession; mucogingival surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2PRF+CAF (Experimental): Two tubes of blood samples were centrifuged by PC-02 Centrifuged device. This centrifuged device is used with 2700 rpm and for 12 minutes( PC-02 Centrifuge, Process,France). PRF were prepared for patients in 2 layer platelet rich fibrin membrane with coronally advanced flap group (2PRF+CAF).
  Following this, in test groups, a horizontal sulcular incision was designed at the buccal side of recession area at the level of CEJ. The incision was extended in the interdental area to be connecting CEJ. The root was planned and hard accumulations were removed but no chemical root treatment was performed. In 2PRF+CAF group: two layers of stacked PRF membranes were positioned over the recession area at the level of CEJ and flpa is positioned coronally.
  Interventions: Device: PC-02 Centrifuge device,2PRF+CAF; Device: PC-02 Centrifuge device, 4 PRF+CAF; Procedure: CTG+CAF
- 4PRF+CAF (Experimental): Four tubes of blood samples were centrifuged by PC-02 Centrifuged device,four layers of PRF membranes were prepared for patients in 4 layer platelet rich fibrin membrane with coronally advanced flap.(4PRF+CAF). This centrifuged device is used with 2700 rpm and for 12 minutes( PC-02 Centrifuge, Process,France) Following this, in test groups, a horizontal sulcular incision was designed at the buccal side of recession area at the level of CEJ. The incision was extended in the interdental area to be connecting CEJ. The root was planned and hard accumulations were removed but no chemical root treatment was performed. In 4PRF+CAF group: four layers of stacked PRF membranes were positioned over the recession area at the level of CEJ and flap is coronally positioned.
  Interventions: Device: PC-02 Centrifuge device,2PRF+CAF; Device: PC-02 Centrifuge device, 4 PRF+CAF; Procedure: CTG+CAF
- CTG+CAF (Active Comparator): The surgical technique in coronally advanced flap with subepithelial connective tissue graft (CTG+CAF) group was "envelope technique" as described by Raetzke. The papillae were dis epithelialized. The root was planned and hard accumulations were removed but no chemical root treatment was performed. The connective tissue graft was harvested from the palate using "trap-door technique" described by Edel. Epithelial layer was elevated with a horizontal and two vertical incisions. The connective tissue graft was harvested as 1 mm by using a standard caliper, then epithelial layer was sutured by resorbable suture. The connective tissue graft was sutured to the recipient bed by resorbable suture at the level of CEJ.
  Interventions: Device: PC-02 Centrifuge device,2PRF+CAF; Device: PC-02 Centrifuge device, 4 PRF+CAF; Procedure: CTG+CAF

INTERVENTIONS:
Device: PC-02 Centrifuge device,2PRF+CAF — In 2PRF+CAF group two layers of stacked PRF membranes were positioned over the recession area at the level of cemento-enamel junction(CEJ). In CAF+2PRF group,two layers of stacked PRF membranes were positioned over the recession area at the level of CEJ
  Other Names: 2 layers Platelet rich fibrin+ coronally advanced flap
Device: PC-02 Centrifuge device, 4 PRF+CAF — Following this, in test groups, a horizontal sulcular incision was designed at the buccal side of recession area at the level of CEJ. The incision was extended in the interdental area to be connecting CEJ. A split thickness flap was raised without vertical incision.18 The papillae were disepithelialized. The root was planned and hard accumulations were removed but no chemical root treatment was performed. In test group-1, two layers of stacked PRF membranes were positioned over the recession area at the level of CEJ. In test group-2, four layers of stacked PRF membranes were positioned over the recession area at the level of CEJ (Figure 2). Membranes were sutured to the recipient bed by a resorbable suture (polyglycolic acid 6/0, Doğsan, Turkey) at the level of CEJ.
  Other Names: 4 layers Platelet Rich Fibrin + coronally advanced flap
Procedure: CTG+CAF — The connective tissue graft was sutured to the recipient bed by resorbable suture at the level of CEJ. Split thickness flap was coronally advanced and sutured by resorbable suture. Finally, periodontal dressing was fixed on the recipient surgical area.
  Other Names: Connective Tissue Graft + Coronally Advanced Flap

SUMMARY:
Miller Class I Gingival Recessions (GR) have been treated by using Coronally Advanced Flap (CAF) with Platelet Rich Fibrin membrane (PRF membrane) or Connective Tissue Graft (CTG). The aim of this study was to evaluate the effect of different multiple layers of PRF membranes for the treatment of GR and compare the results with CTG procedure.

DETAILED DESCRIPTION:
The Coronally Advanced Flap (CAF) has been used in combination with various techniques to increase the coverage and obtain the CRC. CAF+connective tissue graft and CAF+platelet concentrated graft are some of these procedures.

Because of a high success rate in the treatment of GR, CAF combined Connective Tissue Graft (CTG) procedure (bilaminar technique) is considered the gold standard for Miller Class I and II recession defects. According to recent studies CAF + CTG is described as a successful technique with a high CRC value and the percent root coverage achieved with this technique ranges from 79.9% to 89.6%. The advantage of this technique is the enhancement of keratinized tissue width which can be explained by the determination of surface epithelium characteristics of CTG. Moreover, there are disadvantages such as patient's discomfort because of postoperative pain or bleeding and second surgical area.

Therefore, the aim of this study was to evaluate the different doses of PRF membranes for the treatment of Miller Class I gingival recessions and compare with CTG procedure that is considered the gold standard.

MATERIALS AND METHODS In this study, sixty-three Miller Class I gingival recessions in twenty two subjects (10 males and 12 females, aged 21 to 52 years) were treated.

Study design This study was a randomized, controlled clinical trial, with a parallel design comparing different amount layers of PRF membranes and CTG for the treatment of Miller Class I gingival recessions. In the test group-1, 21 randomly selected GR were treated with 2 layers PRF membranes(2PRF)+CAF; in the test group-2, 21 randomly selected GR were treated with 4 layers PRF membranes (4PRF) +CAF and in the control group 21 randomly selected GR were treated with CTG+CAF.

Randomization Subjects were defined to one of the three groups with the use of computer-generated randomization scheme. Allocation concealment was obtained with number labeled opaque envelopes that were opened just before the surgery.

Sample size A software program‡ was used to calculate sample size. The power was calculated 85% when there was 20 gingival recession per each group, using the α value as 0.05.

Clinical measurements All clinical measurements were carried out by one of the examiners. Individual acrylic stents were prepared for all patients to take measurements on the constant points. The following clinical measurements were taken 1 week before surgery (baseline) and at the 1, 3 and 6 months follow up visits: 1) Recession Depth(RD) 2) Recession Width(RW) 3) Keratinized Tissue Height (KTH) 4) Plaque Index(PI), 5) Gingival Index(GI), 6) Probing Depth(PD), 7) Keratinized Tissue Thickness(KTT) 8) Clinical Attachment Level(CAL), 9) Root Coverage(RC). Post operative discomfort and bleeding were recorded using a visual analogue scale (VAS).

Surgical Procedure All surgical operations were performed by the same examiner. Patients received local anesthesia at recession sites and donor sites in the control group. Chlorhexidine mouthwash was performed for intraoral disinfection and antiseptic solution for extraoral disinfection.

Before the surgery, intravenous blood samples were collected from the test group patients. Samples were centrifuged and PRF clots were obtained according to the procedure described by Choukroun.14, 17 Two tubes of blood samples were collected and two layers of PRF membranes were prepared for patients in . Four tubes of blood samples were collected and four layers of PRF membranes were prepared for patients in 4PRF+CAF.

Following this, in test groups, a horizontal sulcular incision was designed at the buccal side of recession area at the level of CEJ. The incision was extended in the interdental area to be connecting CEJ. A split thickness flap was raised without vertical incision. The papillae were disepithelialized. The root was planned and hard accumulations were removed but no chemical root treatment was performed. In 2PRF+CAF group, two layers of stacked PRF membranes were positioned over the recession area at the level of CEJ . In 4PRF+CAF group, four layers of stacked PRF membranes were positioned over the recession area at the level of CEJ. Membranes were sutured to the recipient bed by a 6.0 resorbable suture at the level of CEJ. Split thickness flap was coronally advanced and sutured by a 5.0 resorbable suture.

ELIGIBILITY:
Inclusion Criteria:

1. Periodontally and systemically healthy patient, ≥ 18 years.
2. Miller Class I gingival recession at the buccal aspect of lower and upper incisors, canines or premolars.
3. The presence of ≥ 2 mm keratinized tissue apical to the recession.
4. The presence of identifiable cemento enamel junction (CEJ).
5. ≤ 2 mm probing depth (PD)

Exclusion Criteria:

1. Smoking
2. Pregnancy
3. Periodontal surgery in the past six months.
4. Caries, deep abrasion, restoration or pulpal pathology on the involved tooth.

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline clinical measurement of gingival depth and gingival recession by periodontal Williams Type Probe as millimeter at postoperative 6 month | before surgery and following surgery sixth month
  All clinical measurement were recorded by same periodontal probe(Williams Probe)as height in meters. All measurement were calculated as mean ± standard deviation for per tooth. Clinical measurement following as: 1) Recession Depth: the distance from the CEJ to the most apical point of free gingival margin. 2) Recession Width: horizontal distance of recession in the mesio-distal direction at CEJ 3) Keratinized Tissue Height (KTH): the distance from the mucogingival junction to free gingival margin. 4)Probing Depth 5) Clinical Attachment Level
Change from baseline measurement of keratinized tissue thickness on defects region by spreader and digital calliper at 6 months | before surgery and following surgery sixth month
  2) Keratinized Tissue Thickness (KTT): Keratinized tissue thickness was measured under local anesthesia from a mid-point location between the gingival margin and mucogingival junction with a spreader and its stopper silicon
Change from baseline measurement root coverage at 6 months in millimeters by periodontal probe and change from baseline measurement of root coverage percentage using calculate formula at 6 months | before surgery and following surgery sixth month
  Root Coverage: (RC) was calculated in millimeters and percentages according to the following formulas: [(pre operative RD - post operative RD) / pre operative RD]×100.

SECONDARY OUTCOMES:
Number of participant with treatment related postoperative pain using Visual Analogue Scale on application of PRF and CAF+CTG | first and seventh day
  Post operative discomfort and bleeding were recorded using a visual analogue scale (VAS). The patients enrolled their pain level for the first 7 days after surgery on a horizontal scale, left endpoint means no pain (0), the middle point means pain (50), right endpoint means severe pain (100). Also, patients enrolled the amount of analgesic they used after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rana Culhaoglu, PhD Dr, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan such as share participant individual data. If necessary, then information can be shared.

REFERENCES:
- [Result] Eren G, Atilla G. Platelet-rich fibrin in the treatment of localized gingival recessions: a split-mouth randomized clinical trial. Clin Oral Investig. 2014 Nov;18(8):1941-8. doi: 10.1007/s00784-013-1170-5. Epub 2013 Dec 22. PMID 24362634
- [Result] Keceli HG, Kamak G, Erdemir EO, Evginer MS, Dolgun A. The Adjunctive Effect of Platelet-Rich Fibrin to Connective Tissue Graft in the Treatment of Buccal Recession Defects: Results of a Randomized, Parallel-Group Controlled Trial. J Periodontol. 2015 Nov;86(11):1221-30. doi: 10.1902/jop.2015.150015. Epub 2015 Jul 16. PMID 26177630
- [Result] Tunaliota M, Ozdemir H, Arabaciota T, Gurbuzer B, Pikdoken L, Firatli E. Clinical evaluation of autologous platelet-rich fibrin in the treatment of multiple adjacent gingival recession defects: a 12-month study. Int J Periodontics Restorative Dent. 2015 Jan-Feb;35(1):105-14. doi: 10.11607/prd.1826. PMID 25734713
- [Derived] Culhaoglu R, Taner L, Guler B. Evaluation of the effect of dose-dependent platelet-rich fibrin membrane on treatment of gingival recession: a randomized, controlled clinical trial. J Appl Oral Sci. 2018 May 14;26:e20170278. doi: 10.1590/1678-7757-2017-0278. PMID 29768524